CLINICAL TRIAL: NCT02083939
Title: Prophylactic Antibiotic Treatment for Laparoscopic Inguinal Hernia Mesh Repair: Necessary or Not?
Status: Terminated | Type: Observational
Why Stopped: Recruitment failed
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Danny Rosin, MD, Attending Surgeon, Sheba Medical Center
Other Study IDs: SHEBA-12-9550-DR-CTIL
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Hernia, Inguinal
Keywords: Inguinal hernia; Mesh repair; Prophylactic Antibiotics; Herniorrhaphy; Laparoscopic Inguinal Hernia Repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Antibiotic Prophylaxis: This cohort will receive antibiotic prophylaxis prior to the hernia repair
- No Antibiotic Prophylaxis: This cohort will not receive antibiotic prophylaxis prior to the surgery

SUMMARY:
The purpose of this study is to find out whether it is necessary to prophylactically treat patients undergoing laparoscopic inguinal hernia repairs with antibiotics. Our hypothesis is that it is not necessary to pretreat patients with antibiotics if the operation is minimally invasive with a mesh placed at the defect.

DETAILED DESCRIPTION:
The investigators plan to follow up at least 100 patients who did not receive antibiotics prior to their inguinal hernia repair and compare their outcome to 100 patients who did receive prophylaxis. The investigators mainly will be analyzing the incidence of surgical site infections as evidenced by swelling, redness, pain, warmth or other signs deemed by the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic inguinal hernia repair, unilateral or bilateral

Exclusion Criteria:

* Those requiring antibiotics for the surgery;
* Those patients who have experienced surgical site infections from previous surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients undergoing elective hernia repair will be assigned randomly to the control group; 100 patients will be assigned to the treatment group.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-03; Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection | One year post-operation
  The investigators will interview the patient at one week, at one month, and at one year post-operation and assess for any signs of infection around the location of hernia repair.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Rosin, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Cabaluna ND, Uy GB, Galicia RM, Cortez SC, Yray MD, Buckley BS. A randomized, double-blinded placebo-controlled clinical trial of the routine use of preoperative antibiotic prophylaxis in modified radical mastectomy. World J Surg. 2013 Jan;37(1):59-66. doi: 10.1007/s00268-012-1816-5. PMID 23052809
- [Background] Shah JN, Maharjan SB, Paudyal S. Routine use of antibiotic prophylaxis in low-risk laparoscopic cholecystectomy is unnecessary: a randomized clinical trial. Asian J Surg. 2012 Oct;35(4):136-9. doi: 10.1016/j.asjsur.2012.06.011. Epub 2012 Aug 22. PMID 23063084
- [Background] Wang J, Ji G, Yang Z, Xi M, Wu Y, Zhao P, Wang L, Yu W, Wen A. Prospective randomized, double-blind, placebo controlled trial to evaluate infection prevention in adult patients after tension-free inguinal hernia repair. Int J Clin Pharmacol Ther. 2013 Dec;51(12):924-31. doi: 10.5414/CP201877. PMID 24120711